CLINICAL TRIAL: NCT04204551
Title: Effect of High Intensity Interval Training on Mechanisms of Neuroplasticity and Psychomotor Behaviours in Parkinson's Disease Patients: a Randomized Study With 1-year Follow up
Brief Title: Effect of High Intensity Interval Training on Mechanisms of Neuroplasticity in Parkinson's Disease Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wroclaw University of Health and Sport Sciences (Other)
Collaborators: Józef Piłsudski University of Physical Education (Other); Medical University of Warsaw (Other); Polish Academy of Sciences (Other); Wroclaw Medical University (Other); Military Institute od Medicine National Research Institute (Other)
Responsible Party: Principal Investigator, Jaroslaw Marusiak, Principal Investigator, Wroclaw University of Health and Sport Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017/25/B/NZ7/02795
Record Dates: First submitted 2019-12-04; First posted 2019-12-19 (Actual); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: Parkinson's Disease; Physical Activity; Neurorehabilitation; Neuroplasticity
Keywords: Parkinson's Disease; Physical Activity; Neurorehabilitation; Neuroplasticity; Motor Function; Cognitive Function; Neuroimaging
MeSH Terms: conditions — Parkinson Disease; Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PD-TR (Experimental): Intervention
  exercise, dose: two cycles of 12-week HIIT program (three times a week) separated with 3 months break
  & conventional physical therapy
  Interventions: Behavioral: high-intensity interval training (HIIT); Behavioral: conventional physical therapy
- PD-NTR (Active Comparator): conventional physical therapy
  Interventions: Behavioral: conventional physical therapy
- Healthy Controls (No Intervention): healthy controls without any kind of therapy

INTERVENTIONS:
Behavioral: high-intensity interval training (HIIT) — Two 12-week HIIT cycles will be divided with 3 months of break. Each HIIT cycle will consist of three 1-hour training sessions weekly. Each 1-hour training session will consist of 10-minutes warm-up (at slow voluntary speed), 40-minutes of interval exercise and 10-minutes cool-down phase. The interval exercise part will consist of 10 sets of 4 minutes interval including 2-minutes cycling at ≥ 60 [rpm], but preferably at 80-90 [rpm] (fast phase of interval) and 2-minutes cycling at ≤ 60 [rpm] (slow phase of interval). The training will be performed on a stationary cycle ergometer (MONARK, Ergomedic 874E, Sweden). The heart rate (HR, [bpm]) will be measured by Polar system (Polar, Finland). The patients will pedal on the cycloergometer at 60%-80% of their individualized HRmax.
  Arms: PD-TR
Behavioral: conventional physical therapy — Conventional physical therapy as prescribed and provided by the National Health Fund of Poland, which includes activities for improving motor control, but without any kind of moderate or high intensity aerobic interval or continuous physical training (example: cycle ergometer, treadmill, or Nordic walking training)
  Arms: PD-NTR; PD-TR

SUMMARY:
There are experimental evidences of the important role of high intensity physical exercise in Parkinson's disease (PD) treatment, that induces similar effects to pharmacotherapy. So far, the mechanisms of the impact of these changes on the brain subcortical and cortical regions functioning, motor activities and cognitive functions are still not clear.

The aim of this longitudinal (prospective) human experiment is to examine the effects of two cycles of 12-weeks high-intensity interval training (HIIT) on: (i) the level of dopamine (DA) in putamen in striatum, (ii) neurophysiological function of subcortical and cortical motor structures and skeletal muscle activity, (iii) psychomotor behaviors critically associated with dopamine dependent neural structures functioning and (iv) neurotrophic factors' secretion level in blood.

The investigators will recruit 40 PD individuals, who will be divided into two groups: one of them will perform two 12-weeks cycles of HIIT (PD-TR), and the other will not be trained (PD-NTR) with HIIT. The investigators will also recruit 20 age-matched healthy controls (H-CO) as additional control group who will not perform the HIIT. The PD-TR group will perform the two 12-weeks cycles of the HIIT, that induces beneficial, neuroplastic changes and alleviates the PD symptoms, what was found in earlier studies. All PD subjects (PD-TR and PD-NTR) will be examined during their medication "OFF-phase" (it means after dopaminergic drugs withdrawal) before (Pre) and after (Post) training cycles (first training cycle - HIIT 1; second training cycle - HIIT 2), and namely: Pre HIIT 1, 1 week-, 1.5 month- and 3 months-Post HIIT 1; and then similarly 1 week-, 1.5 month- and 3 months-Post HIIT 2. The subject from H-CO will be tested only once.

To examine the assumed HIIT-induced changes in brain functioning the investigators will apply: (i) the positron emission tomography (PET), (ii) the functional magnetic resonance imaging (fMRI), (iii) electroencephalography (EEG) and (iv) an analysis of neurotrophic factors secretion level in blood. The investigators will also assess motor and non-motor symptoms of PD and psychomotor behaviors based on neuropsychological tests of cognitive functions and manual dexterity.

The results of this project will help to answer the fundamental questions about HIIT induced mechanisms of neuroplasticity in PD patients, what is important from scientific and treatment-strategy point of view.

DETAILED DESCRIPTION:
I. Research Project Objectives

Aim 1. To examine the effect of two HIIT cycles on presynaptic striatal DA availability (in dorsal putamen) in the tested PD patients using PET imaging method with the 18F-dopa - [18F]fluorodopa uptake, which provides in this case a very good index of restored striatal presynaptic dopaminergic function (Brooks and Pavese, 2011).

Hypothesis 1. The presynaptic striatal dopaminergic function will improve (18F-dopa uptake increase) after the first and second bout of HIIT cycle compared to baseline in the PD-TR group, and will sustain in 1 year follow up time frame (3 months after the second HIIT cycle cessation). In the PD-NTR group, the presynaptic striatal dopaminergic function will not improve or even will be worsened (18F-dopa uptake decrease) in the same time interval. Importantly for this hypothesis the annual decrease of putaminal 18F-dopa is about 10% in early PD (Morrish et al., 1995).

Aim 2. To characterize an influence of two HIIT cycles on neurophysiological functions (NPFs) of: (i) motor and cognitive subcortical and cortical structures, (that are critically dependant on the presynaptic DA availability), using fMRI and EEG, and (ii) skeletal muscles engaged in motor task, using surface EMG. The following neurophysiological functions of central nervous system (CNS) will be tested during performance of the DA availability-dependant self initiated index finger motor task and during mental imagery of this motor task (cognitive task): (i) a level of activation of subcortical and cortical structures, and (ii) strength of functional coupling (functional connectivity) between neural structures. For skeletal muscles NPFs', the investigators will study a strategy of motor units activation. Also, since the investigators will record EEG and EMG simultaneously, the investigators will assess strength of cortico-muscular coupling.

Hypothesis 2. NPFs will improve after the first and second bout of HIIT cycle compared to baseline in the PD-TR group, and will sustain in 1 year follow up time frame. Namely, the investigators speculate that for the motor task and mental imagery task in CNS activity, it will be: (1) an increase of activation in substantia nigra (SN), putamen (PUT), primary motor cortex (M1), supplementary motor area (SMA); (2) decrease of activation of lateral premotor cortex (PMC) and cerebellum; with simultaneous (3) increase of functional coupling of: SN with PUT; PUT with M1, PMC, SMA and dorsolateral prefrontal cortex (DLPFC); and DLPFC with M1, PMC, SMA and cerebellum; (4) decrease of functional coupling between M1, PMC, SMA, cerebellum and parietal cortex; and (5) for the mental imagery task the investigators additionally assume an increase of parietal and decrease of occipital cortex activation. For the skeletal muscle function it will be an improvement in recruitment strategy of motor units. Taking into the data from the simultaneous recording of electrical activity of brain cortex and skeletal muscles engaged in motor tasks, the investigators assume strengthening of corticomuscular coupling. In the PD-NTR group NPFs will not improve or even will be worsened in the same time interval and especially after the 1 year from the baseline.

Aim 3. To characterize an influence of two HIIT cycles on the psychomotor behaviors (PMBs), critically dependant on the DA availability and brain's NPFs. The following PMBs will be tested during several experiments: (1) self initiated bimanual anti-phase index finger flexion/extension movement task and mental imagery of this task during the fMRI scans, (2) self initiated bimanual anti-phase index finger abduction/adduction movement task and mental imagery of this task during the simultaneous EEG, EMG and force recordings; (3) simple functional test of bimanual dexterity (using peg board test), (4) all motor and non-motor PD symptoms evaluation, based on neurological assessment, (5) overall cognitive function and specifically aspects of executive function using psychological tests.

Hypothesis 3. PMBs will improve after the first and second bout of HIIT cycle compared to baseline in the PD-TR group, and will sustain in 1 year follow up time frame, as a consequence of the improvements of presynaptic striatal DA availability and NPFs, The PMBs improvement will not be present in the PD-NTR group, or even the PMBs will be worsened in the same time interval and especially after the 1 year from the baseline.

Aim 4. To evaluate: (i) the effect of two HIIT cycles on BDNF (brain-derived neurotrophic factor), NGF (nerve growth factor), IGF-1 (insulin like growth factor type 1) secretion level in blood treated as markers of neuroplasticity efficiency and (ii) an influence of BDNF polymorphism on PD patients neuroplastic responsiveness to HIIT (expressed in exercise-induced increase of presynaptic DA level, and improvement of NPF' and PMBs).

Hypothesis 4. The secretion level of the BDNF, NGF and IGF-1 will increase after the first and second bout of HIIT cycle compared to baseline in the PD-TR group, and will sustain in 1 year follow up time frame. In contrary to PD-TR group, the improvement in BDNF, NGF and IGF-1 secretion level will not be present in the PD-NTR group or even their level will decrease after 1 year follow up. The PD patients neuroplastic responsiveness to HIIT will be influenced by the BDNF polymorphism type, with potentially worse responsiveness for the Val66Met polymorphism of BDNF (this polymorphism causes a valine to methionine change at position 66 of the proBDNF protein).

Aim 5. To investigate the relationships of presynaptic DA availability with the NPFs, PMBs and BDNF level of specific polymorphism type.

Hypothesis 5. The investigators hypothesize that, the HIIT related increase of presynaptic DA availability will be significantly positively correlated with: (i) an improvement of NPFs and PMBs, and with an increased level of BDNF secretion in blood, and (ii) negatively with the BDNF Val66Met polymorphism type in PD-TR group. Contrary to the above, there will be lack or less significant correlations of presynaptic striatal DA availability with NPFs, PMBs and BDNF level in the PD-NTR group.

II. Research design and work plan

This project is a longitudinal, 1-year follow up randomized controlled study with 3 arms. Whole block type randomization process is carried out by the investigators of this study using sequentially numbered sealed envelopes. Opaque envelopes are used to conceal allocation. The project enrolls two PD patients' groups: PD-TR - the PD patients who will perform physical training cycle; PD-NTR - non-trained PD patients and one H-CO - healthy control group that will not perform the HIIT cycles. All PD subjects (PD-TR and PD-NTR) will be examined during their medication "OFF-phase" in the following time points: Pre HIIT 1, 1 week-, 1.5 month- and 3 months-Post HIIT 1; and then similarly 1 week-, 1.5 month- and 3 months-Post HIIT 2. The subject from H-CO will be tested only once.

III. Research methodology

III.1.1. Subjects characteristics The 40 PD individuals (aged 45-65 years), are qualified to the study after being diagnosed to have an idiopathic PD, based on neurological assessment. The diagnosis of Parkinson's disease are based on medical history, physical and neurological examinations and response to L-dopa. Patients are clinically assessed with the UPDRS and the H&Y scale by experienced movement disorder neurologist. To obtain the most homogeneous group of patients with unified type of medication (important for PET measurements), that will be able to perform HIIT cycle and participate fully in the testing sessions, the investigators limit patients' recruitment to mild PD (1-2 points in H&Y scale) with prevalence of bradykinesia and absence or less accentuated tremor. The healthy control group will comprise of age-, gender, height- and body mass-matched healthy individuals.

III.1.2. Subjects recruitment The PD subjects are recruited from Neurology Clinics in Warsaw, Poland. The healthy elderly control group of subjects are recruited based on: (i) public advertisement and (ii) contacts with the Universities of the Third Age and the Seniors' Clubs around the Warsaw city.

III.2. Training procedures The patients from PD-TR group will perform two 12-week HIIT cycles divided with 3 months of break. This HIIT cycle will consist of three 1-hour training sessions weekly. Each 1-hour training session will consist of 10-minutes warm-up (at slow voluntary speed), 40-minutes of interval exercise and 10-minutes cool-down phase. In each training session, the interval exercise part will consist of 10 sets of 4 minutes interval including 2-minutes cycling at ≥ 60 [rpm], but preferably at 80-90 [rpm] (fast phase of interval) and 2-minutes cycling at ≤ 60 [rpm] (slow phase of interval). The training will be performed on a stationary cycle ergometer (MONARK, Ergomedic 874E, Sweden), that allows to measure cadence [rpm]) and power [W]. The heart rate (HR, [bpm]) will be measured by Polar system (Polar, Finland). Training supervisor will adjust the resistance for each patient to ensure cycling at each patient's target heart rate (THR) and with appropriate speed. All training sessions will be performed while the patients' medication on-phase (beneficial effect of anti-parkinsonian medication). The patients will pedal on the cycloergometer at 60%-80% of their individualized HRmax and will be encouraged to cycle faster (80-90 rpm, or 30% faster than their preferred voluntary speed) during the fast phase of the interval training. Each patient will increased his/her target heart rate every 2 weeks by 5% from 60% up to 80% in the following order: 60% of the HRmax during the first two weeks, 65% during the 3-4 week, 70% during 5-6 week, 75% during 7-9 week and 80% during 10-12 week of training period. During each part of these 36 training sessions (warm up; fast and slow phase of interval training part; slow down), for each subject, the investigators will measure: (i) the values of the % of HRmax, (ii) cadence and power, and (iii) patients' perception of exercise intensity using the Borg Rating of Perceived Exertion (RPE) (Borg, 1982). To enhance the cognitive engagement in exercised PD patients the cadence (cycling speed) data will be presented on each patient's screen using custom-made feedback system. The patient will see two vertical bars, on which the first is going to be the set target level of speed (appropriate for the slow or fast phase of interval) and the second is going to be the an actual speed generated by exercising patient. Additionally, the PD patients will be cued with metronome and verbal comments of instructor to pedal with appropriate rhythm which will be adjusted to the set speed.

IV. Statistical analysis

The investigators will first perform a between-group comparison for all demographics and clinical characteristics to check for baseline differences (Student's t test or Mann-Whitney U tests for normally and non-normally distributed data or the Fisher's exact test for contingency data). Repeated measures ANOVA will be used to perform a between-group comparison of changes in the testing points. Significant main effects will then be subjected to a post-hoc pair-wise comparison primarily between PD-TR and PD-NTR, and PD-TR and H-CO. Correlation analysis (Pearson or Spearman correlation coefficient) will be performed between PET data (showing DA availability), and fMRI, EEG, EMG (describing NPFs), PMBs, and neuroplasticity markers outcomes. For all analyses, a significance level will be set to α=0.05 with Bonferroni adjustments for multiple comparisons when necessary.

ELIGIBILITY:
Inclusion Criteria:

* for PD patients: age 45-65 years-old; diagnosis of idiopathic PD; and modified Hoehn and Yahr stages between 1.5 and 3
* for healthy controls: age-matched to PD patients, lack of neurological disorders
* all participants will also satisfy the following eligibility criteria: (i) proficient in Polish; (ii) no significant cognitive impairments (dementia), as assessed by the MMSE test (Folstein et al., 1975) score ≥ 27; (iii) no prior history of neurological, psychiatric, or other disorders that may influence CNS structure and function; (iv) no current medication to affect cognitive psychomotor functioning (opioid analgesics, anxiolytics or antidepressants) and (v) signed informed consent.

Exclusion Criteria:

* for PD patients: (1) presence of other neurological disorders, (2) any cardiovascular and respiratory system restrictions and/or motor deficits that could limit performance in high-speed pedaling on a cycle ergometer or in the conventional physical therapy and (3) practicing any regular intensive physical activity except for physical therapy for PD
* for healthy controls: presence of neurological disorders
* for all tested subjects, an additional exclusion criterion for the PET and fMRI experiments will be a claustrophobia.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-02-15 (Actual); Primary Completion 2020-09-25 (Estimated); Study Completion 2020-12-18 (Estimated)

PRIMARY OUTCOMES:
Positron Emission Tomography (PET) with 18F-dopa - PET imaging with [18F]fluorodopa uptake. | Pre-HIIT 1 - it means up to 1-week before the HIIT 1 starts
  To examine presynaptic striatal DA availability (in dorsal putamen) using PET imaging method with the 18F-dopa - [18F]fluorodopa uptake. The recordings will be expressed in Ki ref values [Ki ref] and Standard Uptake Values [SUV].
Positron Emission Tomography (PET) with 18F-dopa - PET imaging with [18F]fluorodopa uptake. | 1-week Post-HIIT 1
  To examine presynaptic striatal DA availability (in dorsal putamen) using PET imaging method with the 18F-dopa - [18F]fluorodopa uptake. The recordings will be expressed in Ki ref values [Ki ref] and Standard Uptake Values [SUV].
Positron Emission Tomography (PET) with 18F-dopa - PET imaging with [18F]fluorodopa uptake. | 3-months Post-HIIT 2
  To examine presynaptic striatal DA availability (in dorsal putamen) using PET imaging method with the 18F-dopa - [18F]fluorodopa uptake. The recordings will be expressed in Ki ref values [Ki ref] and Standard Uptake Values [SUV].
functional Magnetic Resonance Imaging (fMRI) - metabolic activity of brain recorded with MRI scanner. | Pre-HIIT 1 - it means up to 1-week before the HIIT 1 starts
  To evaluate neurophysiological functions of brain subcortical and cortical structures using MRI scanner. The recordings will be conducted at rest and during self initiated index finger motor task and during mental imagery of this motor task. The image recordings will express metabolic brain activity as expressed in fMRI response [% BOLD signal].
functional Magnetic Resonance Imaging (fMRI) - metabolic activity of brain recorded with MRI scanner. | 1-week Post-HIIT 1
  To evaluate neurophysiological functions of brain subcortical and cortical structures using MRI scanner. The recordings will be conducted at rest and during self initiated index finger motor task and during mental imagery of this motor task. The image recordings will express metabolic brain activity as expressed in fMRI response [% BOLD signal].
functional Magnetic Resonance Imaging (fMRI) - metabolic activity of brain recorded with MRI scanner. | 3-months Post-HIIT 2
  To evaluate neurophysiological functions of brain subcortical and cortical structures using MRI scanner. The recordings will be conducted at rest and during self initiated index finger motor task and during mental imagery of this motor task. The image recordings will express metabolic brain activity as expressed in fMRI response [% BOLD signal].
Electroencephalography (EEG) - amplitude of EEG event related potentials of brain cortex recorded from scalp using surface electrodes. | Pre-HIIT 1 - it means up to 1-week before the HIIT1 starts
  To evaluate neurophysiological functions of brain cortical structures, electroencephalography (EEG - electrical activity of brain cortex) will be recorded from scalp using 128-chanel system. The recordings will be conducted at rest and during self initiated index finger motor task and during mental imagery of this motor task. The recordings will be analyzed as an amplitude of event related potentials and expressed in microvolts [µV].
Electroencephalography (EEG) - amplitude of EEG event related potentials of brain cortex recorded from scalp using surface electrodes. | 1-week Post-HIIT 1
  To evaluate neurophysiological functions of brain cortical structures, electroencephalography (EEG - electrical activity of brain cortex) will be recorded from scalp using 128-chanel system. The recordings will be conducted at rest and during self initiated index finger motor task and during mental imagery of this motor task. The recordings will be analyzed as an amplitude of event related potentials and expressed in microvolts [µV].
Electroencephalography (EEG) - amplitude of EEG event related potentials of brain cortex recorded from scalp using surface electrodes. | 1.5-month Post-HIIT 1
  To evaluate neurophysiological functions of brain cortical structures, electroencephalography (EEG - electrical activity of brain cortex) will be recorded from scalp using 128-chanel system. The recordings will be conducted at rest and during self initiated index finger motor task and during mental imagery of this motor task. The recordings will be analyzed as an amplitude of event related potentials and expressed in microvolts [µV].
Electroencephalography (EEG) - amplitude of EEG event related potentials of brain cortex recorded from scalp using surface electrodes. | 3-months Post-HIIT 1
  To evaluate neurophysiological functions of brain cortical structures, electroencephalography (EEG - electrical activity of brain cortex) will be recorded from scalp using 128-chanel system. The recordings will be conducted at rest and during self initiated index finger motor task and during mental imagery of this motor task. The recordings will be analyzed as an amplitude of event related potentials and expressed in microvolts [µV].
Electroencephalography (EEG) - amplitude of EEG event related potentials of brain cortex recorded from scalp using surface electrodes. | 1-week Post-HIIT 2
  To evaluate neurophysiological functions of brain cortical structures, electroencephalography (EEG - electrical activity of brain cortex) will be recorded from scalp using 128-chanel system. The recordings will be conducted at rest and during self initiated index finger motor task and during mental imagery of this motor task. The recordings will be analyzed as an amplitude of event related potentials and expressed in microvolts [µV].
Electroencephalography (EEG) - amplitude of EEG event related potentials of brain cortex recorded from scalp using surface electrodes. | 1.5-month Post-HIIT 2
  To evaluate neurophysiological functions of brain cortical structures, electroencephalography (EEG - electrical activity of brain cortex) will be recorded from scalp using 128-chanel system. The recordings will be conducted at rest and during self initiated index finger motor task and during mental imagery of this motor task. The recordings will be analyzed as an amplitude of event related potentials and expressed in microvolts [µV].
Electroencephalography (EEG) - amplitude of EEG event related potentials of brain cortex recorded from scalp using surface electrodes. | 3-months Post-HIIT 2
  To evaluate neurophysiological functions of brain cortical structures, electroencephalography (EEG - electrical activity of brain cortex) will be recorded from scalp using 128-chanel system. The recordings will be conducted at rest and during self initiated index finger motor task and during mental imagery of this motor task. The recordings will be analyzed as an amplitude of event related potentials and expressed in microvolts [µV].
Electroencephalography (EEG) - latency of EEG event related potentials of brain cortex recorded from scalp using surface electrodes. | Pre-HIIT 1 - it means up to 1-week before the HIIT1 starts
  To evaluate neurophysiological functions of brain cortical structures, electroencephalography (EEG - electrical activity of brain cortex) will be recorded from scalp using 128-chanel system. The recordings will be conducted at rest and during self initiated index finger motor task and during mental imagery of this motor task. The recordings will be analyzed as a latency of event related potentials and expressed in milliseconds [ms].
Electroencephalography (EEG) - latency of EEG event related potentials of brain cortex recorded from scalp using surface electrodes. | 1-week Post-HIIT 1
  To evaluate neurophysiological functions of brain cortical structures, electroencephalography (EEG - electrical activity of brain cortex) will be recorded from scalp using 128-chanel system. The recordings will be conducted at rest and during self initiated index finger motor task and during mental imagery of this motor task. The recordings will be analyzed as a latency of event related potentials and expressed in milliseconds [ms].
Electroencephalography (EEG) - latency of EEG event related potentials of brain cortex recorded from scalp using surface electrodes. | 1.5-month Post-HIIT 1
  To evaluate neurophysiological functions of brain cortical structures, electroencephalography (EEG - electrical activity of brain cortex) will be recorded from scalp using 128-chanel system. The recordings will be conducted at rest and during self initiated index finger motor task and during mental imagery of this motor task. The recordings will be analyzed as a latency of event related potentials and expressed in milliseconds [ms].
Electroencephalography (EEG) - latency of EEG event related potentials of brain cortex recorded from scalp using surface electrodes. | 3-months Post-HIIT 1
  To evaluate neurophysiological functions of brain cortical structures, electroencephalography (EEG - electrical activity of brain cortex) will be recorded from scalp using 128-chanel system. The recordings will be conducted at rest and during self initiated index finger motor task and during mental imagery of this motor task. The recordings will be analyzed as a latency of event related potentials and expressed in milliseconds [ms].
Electroencephalography (EEG) - latency of EEG event related potentials of brain cortex recorded from scalp using surface electrodes. | 1-week Post-HIIT 2
  To evaluate neurophysiological functions of brain cortical structures, electroencephalography (EEG - electrical activity of brain cortex) will be recorded from scalp using 128-chanel system. The recordings will be conducted at rest and during self initiated index finger motor task and during mental imagery of this motor task. The recordings will be analyzed as a latency of event related potentials and expressed in milliseconds [ms].
Electroencephalography (EEG) - latency of EEG event related potentials of brain cortex recorded from scalp using surface electrodes. | 1.5-month Post-HIIT 2
  To evaluate neurophysiological functions of brain cortical structures, electroencephalography (EEG - electrical activity of brain cortex) will be recorded from scalp using 128-chanel system. The recordings will be conducted at rest and during self initiated index finger motor task and during mental imagery of this motor task. The recordings will be analyzed as a latency of event related potentials and expressed in milliseconds [ms].
Electroencephalography (EEG) - latency of EEG event related potentials of brain cortex recorded from scalp using surface electrodes. | 3-months Post-HIIT 2
  To evaluate neurophysiological functions of brain cortical structures, electroencephalography (EEG - electrical activity of brain cortex) will be recorded from scalp using 128-chanel system. The recordings will be conducted at rest and during self initiated index finger motor task and during mental imagery of this motor task. The recordings will be analyzed as a latency of event related potentials and expressed in milliseconds [ms].
Electroencephalography (EEG) - EEG power in the beta-band recorded from scalp using surface electrodes. | Pre-HIIT 1 - it means up to 1-week before the HIIT1 starts
  To evaluate neurophysiological functions of brain cortical structures, electroencephalography (EEG - electrical activity of brain cortex) will be recorded from scalp using 128-chanel system. The recordings will be conducted at rest and during self initiated index finger motor task and during mental imagery of this motor task. The recordings will be analyzed as the EEG power in the beta-band (≈13-35 Hz) and expressed in decibels [dB].
Electroencephalography (EEG) - EEG power in the beta-band recorded from scalp using surface electrodes. | 1-week Post-HIIT 1
  To evaluate neurophysiological functions of brain cortical structures, electroencephalography (EEG - electrical activity of brain cortex) will be recorded from scalp using 128-chanel system. The recordings will be conducted at rest and during self initiated index finger motor task and during mental imagery of this motor task. The recordings will be analyzed as the EEG power in the beta-band (≈13-35 Hz) and expressed in decibels [dB].
Electroencephalography (EEG) - EEG power in the beta-band recorded from scalp using surface electrodes. | 1.5-month Post-HIIT 1
  To evaluate neurophysiological functions of brain cortical structures, electroencephalography (EEG - electrical activity of brain cortex) will be recorded from scalp using 128-chanel system. The recordings will be conducted at rest and during self initiated index finger motor task and during mental imagery of this motor task. The recordings will be analyzed as the EEG power in the beta-band (≈13-35 Hz) and expressed in decibels [dB].
Electroencephalography (EEG) - EEG power in the beta-band recorded from scalp using surface electrodes. | 3-months Post-HIIT 1
  To evaluate neurophysiological functions of brain cortical structures, electroencephalography (EEG - electrical activity of brain cortex) will be recorded from scalp using 128-chanel system. The recordings will be conducted at rest and during self initiated index finger motor task and during mental imagery of this motor task. The recordings will be analyzed as the EEG power in the beta-band (≈13-35 Hz) and expressed in decibels [dB].
Electroencephalography (EEG) - EEG power in the beta-band recorded from scalp using surface electrodes. | 1-week Post-HIIT 2
  To evaluate neurophysiological functions of brain cortical structures, electroencephalography (EEG - electrical activity of brain cortex) will be recorded from scalp using 128-chanel system. The recordings will be conducted at rest and during self initiated index finger motor task and during mental imagery of this motor task. The recordings will be analyzed as the EEG power in the beta-band (≈13-35 Hz) and expressed in decibels [dB].
Electroencephalography (EEG) - EEG power in the beta-band recorded from scalp using surface electrodes. | 1.5-month Post-HIIT 2
  To evaluate neurophysiological functions of brain cortical structures, electroencephalography (EEG - electrical activity of brain cortex) will be recorded from scalp using 128-chanel system. The recordings will be conducted at rest and during self initiated index finger motor task and during mental imagery of this motor task. The recordings will be analyzed as the EEG power in the beta-band (≈13-35 Hz) and expressed in decibels [dB].
Electroencephalography (EEG) - EEG power in the beta-band recorded from scalp using surface electrodes. | 3-months Post-HIIT 2
  To evaluate neurophysiological functions of brain cortical structures, electroencephalography (EEG - electrical activity of brain cortex) will be recorded from scalp using 128-chanel system. The recordings will be conducted at rest and during self initiated index finger motor task and during mental imagery of this motor task. The recordings will be analyzed as the EEG power in the beta-band (≈13-35 Hz) and expressed in decibels [dB].
Electromyography (EMG) - recordings of electrical activity of skeletal muscles using surface electrodes. | Pre-HIIT 1 - it means up to 1-week before the HIIT 1 starts
  To evaluate neurophysiological functions of muscles engaged in an activity (hand muscles), electromyography (EMG - recordings of electrical activity of skeletal muscles) will be collected using surface electrodes, during index finger motor tasks and at rest. The recordings will be expressed in millivolts [mV].
Electromyography (EMG) - recordings of electrical activity of skeletal muscles using surface electrodes. | 1-week Post-HIIT 1
  To evaluate neurophysiological functions of muscles engaged in an activity (hand muscles), electromyography (EMG - recordings of electrical activity of skeletal muscles) will be collected using surface electrodes, during index finger motor tasks and at rest. The recordings will be expressed in millivolts [mV].
Electromyography (EMG) - recordings of electrical activity of skeletal muscles using surface electrodes. | 1.5-month Post-HIIT 1
  To evaluate neurophysiological functions of muscles engaged in an activity (hand muscles), electromyography (EMG - recordings of electrical activity of skeletal muscles) will be collected using surface electrodes, during index finger motor tasks and at rest. The recordings will be expressed in millivolts [mV].
Electromyography (EMG) - recordings of electrical activity of skeletal muscles using surface electrodes. | 3-months Post-HIIT 1
  To evaluate neurophysiological functions of muscles engaged in an activity (hand muscles), electromyography (EMG - recordings of electrical activity of skeletal muscles) will be collected using surface electrodes, during index finger motor tasks and at rest. The recordings will be expressed in millivolts [mV].
Electromyography (EMG) - recordings of electrical activity of skeletal muscles using surface electrodes. | 1-week Post-HIIT 2
  To evaluate neurophysiological functions of muscles engaged in an activity (hand muscles), electromyography (EMG - recordings of electrical activity of skeletal muscles) will be collected using surface electrodes, during index finger motor tasks and at rest. The recordings will be expressed in millivolts [mV].
Electromyography (EMG) - recordings of electrical activity of skeletal muscles using surface electrodes. | 1.5-month Post-HIIT 2
  To evaluate neurophysiological functions of muscles engaged in an activity (hand muscles), electromyography (EMG - recordings of electrical activity of skeletal muscles) will be collected using surface electrodes, during index finger motor tasks and at rest. The recordings will be expressed in millivolts [mV].
Electromyography (EMG) - recordings of electrical activity of skeletal muscles using surface electrodes. | 3-months Post-HIIT 2
  To evaluate neurophysiological functions of muscles engaged in an activity (hand muscles), electromyography (EMG - recordings of electrical activity of skeletal muscles) will be collected using surface electrodes, during index finger motor tasks and at rest. The recordings will be expressed in millivolts [mV].
Purdue Pegboard Test (PPT) - neuropsychological test | Pre-HIIT 1 - it means up to 1-week before the HIIT 1 starts
  To evaluate executive function and bimanual dexterity. The Purdue Pegboard consists of a test board, score sheets and elements to work with: pins, collars, washers. Subjects are instructed to insert pins to holes in the board or build the sets with the elements in a fixed time. The final score is the number of pins inserted or built sets [number of pins or sets].
Purdue Pegboard Test (PPT) - neuropsychological test | 1-week Post-HIIT 1
  To evaluate executive function and bimanual dexterity. The Purdue Pegboard consists of a test board, score sheets and elements to work with: pins, collars, washers. Subjects are instructed to insert pins to holes in the board or build the sets with the elements in a fixed time. The final score is the number of pins inserted or built sets [number of pins or sets].
Purdue Pegboard Test (PPT) - neuropsychological test | 1.5-month Post-HIIT 1
  To evaluate executive function and bimanual dexterity. The Purdue Pegboard consists of a test board, score sheets and elements to work with: pins, collars, washers. Subjects are instructed to insert pins to holes in the board or build the sets with the elements in a fixed time. The final score is the number of pins inserted or built sets [number of pins or sets].
Purdue Pegboard Test (PPT) - neuropsychological test | 3-months Post-HIIT 1
  To evaluate executive function and bimanual dexterity. The Purdue Pegboard consists of a test board, score sheets and elements to work with: pins, collars, washers. Subjects are instructed to insert pins to holes in the board or build the sets with the elements in a fixed time. The final score is the number of pins inserted or built sets [number of pins or sets].
Purdue Pegboard Test (PPT) - neuropsychological test | 1-week Post-HIIT 2
  To evaluate executive function and bimanual dexterity. The Purdue Pegboard consists of a test board, score sheets and elements to work with: pins, collars, washers. Subjects are instructed to insert pins to holes in the board or build the sets with the elements in a fixed time. The final score is the number of pins inserted or built sets [number of pins or sets].
Purdue Pegboard Test (PPT) - neuropsychological test | 1.5-month Post-HIIT 2
  To evaluate executive function and bimanual dexterity. The Purdue Pegboard consists of a test board, score sheets and elements to work with: pins, collars, washers. Subjects are instructed to insert pins to holes in the board or build the sets with the elements in a fixed time. The final score is the number of pins inserted or built sets [number of pins or sets].
Purdue Pegboard Test (PPT) - neuropsychological test | 3-months Post-HIIT 2
  To evaluate executive function and bimanual dexterity. The Purdue Pegboard consists of a test board, score sheets and elements to work with: pins, collars, washers. Subjects are instructed to insert pins to holes in the board or build the sets with the elements in a fixed time. The final score is the number of pins inserted or built sets [number of pins or sets].
TMT-A - trail making test, part A | Pre-HIIT 1 - it means up to 1-week before the HIIT 1 starts
  TMT-A is a psychological measure of cognitive processing speed, measured as performance time (the shorter the time the better performance), expressed in [s].
TMT-A - trail making test, part A | 1-week Post-HIIT 1
  TMT-A is a psychological measure of cognitive processing speed, measured as performance time (the shorter the time the better performance), expressed in [s].
TMT-A - trail making test, part A | 1.5-month Post-HIIT 1
  TMT-A is a psychological measure of cognitive processing speed, measured as performance time (the shorter the time the better performance), expressed in [s].
TMT-A - trail making test, part A | 3-months Post-HIIT 1
  TMT-A is a psychological measure of cognitive processing speed, measured as performance time (the shorter the time the better performance), expressed in [s].
TMT-A - trail making test, part A | 1-week Post-HIIT 2
  TMT-A is a psychological measure of cognitive processing speed, measured as performance time (the shorter the time the better performance), expressed in [s].
TMT-A - trail making test, part A | 1.5-month Post-HIIT 2
  TMT-A is a psychological measure of cognitive processing speed, measured as performance time (the shorter the time the better performance), expressed in [s].
TMT-A - trail making test, part A | 3-months Post-HIIT 2
  TMT-A is a psychological measure of cognitive processing speed, measured as performance time (the shorter the time the better performance), expressed in [s].
TMT-B - trail making test, part B | Pre-HIIT 1 - it means up to 1-week before the HIIT1 starts
  TMT-B is a psychological measure of executive function, measured as performance time (the shorter the time the better performance), expressed in [s].
TMT-B - trail making test, part B | 1-week Post-HIIT 1
  TMT-B is a psychological measure of executive function, measured as performance time (the shorter the time the better performance), expressed in [s].
TMT-B - trail making test, part B | 1.5-month Post-HIIT 1
  TMT-B is a psychological measure of executive function, measured as performance time (the shorter the time the better performance), expressed in [s].
TMT-B - trail making test, part B | 3-months Post-HIIT 1
  TMT-B is a psychological measure of executive function, measured as performance time (the shorter the time the better performance), expressed in [s].
TMT-B - trail making test, part B | 1-week Post-HIIT 2
  TMT-B is a psychological measure of executive function, measured as performance time (the shorter the time the better performance), expressed in [s].
TMT-B - trail making test, part B | 1.5-month Post-HIIT 2
  TMT-B is a psychological measure of executive function, measured as performance time (the shorter the time the better performance), expressed in [s].
TMT-B - trail making test, part B | 3-months Post-HIIT 2
  TMT-B is a psychological measure of executive function, measured as performance time (the shorter the time the better performance), expressed in [s].
ST-I - Stroop Test, part I | Pre-HIIT 1 - it means up to 1-week before the HIIT 1 starts
  ST-I is used as a psychological measure of processing speed, measured as performance time (the shorter the time the better performance), expressed in [s].
ST-I - Stroop Test, part I | 1-week Post-HIIT 1
  ST-I is used as a psychological measure of processing speed, measured as performance time (the shorter the time the better performance), expressed in [s].
ST-I - Stroop Test, part I | 1.5-month Post-HIIT 1
  ST-I is used as a psychological measure of processing speed, measured as performance time (the shorter the time the better performance), expressed in [s].
ST-I - Stroop Test, part I | 3-months Post-HIIT 1
  ST-I is used as a psychological measure of processing speed, measured as performance time (the shorter the time the better performance), expressed in [s].
ST-I - Stroop Test, part I | 1-week Post-HIIT 2
  ST-I is used as a psychological measure of processing speed, measured as performance time (the shorter the time the better performance), expressed in [s].
ST-I - Stroop Test, part I | 1.5-month Post-HIIT 2
  ST-I is used as a psychological measure of processing speed, measured as performance time (the shorter the time the better performance), expressed in [s].
ST-I - Stroop Test, part I | 3-months Post-HIIT 2
  ST-I is used as a psychological measure of processing speed, measured as performance time (the shorter the time the better performance), expressed in [s].
ST-II - Stroop Test, part II | Pre-HIIT 1 - it means up to 1-week before the HIIT 1 starts
  ST-II is used as a psychological measure of selective attention and inhibition, measured as performance time (the shorter the time the better performance), expressed in [s].
ST-II - Stroop Test, part II | 1-week Post-HIIT 1
  ST-II is used as a psychological measure of selective attention and inhibition, measured as performance time (the shorter the time the better performance), expressed in [s].
ST-II - Stroop Test, part II | 1.5-month Post-HIIT 1
  ST-II is used as a psychological measure of selective attention and inhibition, measured as performance time (the shorter the time the better performance), expressed in [s].
ST-II - Stroop Test, part II | 3-months Post-HIIT 1
  ST-II is used as a psychological measure of selective attention and inhibition, measured as performance time (the shorter the time the better performance), expressed in [s].
ST-II - Stroop Test, part II | 1-week Post-HIIT 2
  ST-II is used as a psychological measure of selective attention and inhibition, measured as performance time (the shorter the time the better performance), expressed in [s].
ST-II - Stroop Test, part II | 1.5-month Post-HIIT 2
  ST-II is used as a psychological measure of selective attention and inhibition, measured as performance time (the shorter the time the better performance), expressed in [s].
ST-II - Stroop Test, part II | 3-months Post-HIIT 2
  ST-II is used as a psychological measure of selective attention and inhibition, measured as performance time (the shorter the time the better performance), expressed in [s].
UPDRS - unified Parkinson's disease rating scale | Pre-HIIT 1 - it means up to 1-week before the HIIT 1 starts
  Motor and non-motor Parkinson's disease signs/symptoms will be evaluated using UPDRS (sections I - III, that include the items 1 -31). Each item is expressed in [points] from 0 to 4 points, with an interpretation that the higher value means the severe accentuation of sign/symptom. The total score will be reported, as the sum of the points of the sections I-III (the score in the range 0 - 176 points) and each section's score will be reported as well, i.e.: the sum of the points of the section I (sum of points for items 1-4 in the range 0 - 16 points), the sum of the points of the section II (sum of points for items 5-17 in the range 0 - 52 points), the sum of the points of the section III (sum of points for items 18-31 in the range 0 - 108 points).
UPDRS - unified Parkinson's disease rating scale | 1-week Post-HIIT 1
  Motor and non-motor Parkinson's disease signs/symptoms will be evaluated using UPDRS (sections I - III, that include the items 1 -31). Each item is expressed in [points] from 0 to 4 points, with an interpretation that the higher value means the severe accentuation of sign/symptom. The total score will be reported, as the sum of the points of the sections I-III (the score in the range 0 - 176 points) and each section's score will be reported as well, i.e.: the sum of the points of the section I (sum of points for items 1-4 in the range 0 - 16 points), the sum of the points of the section II (sum of points for items 5-17 in the range 0 - 52 points), the sum of the points of the section III (sum of points for items 18-31 in the range 0 - 108 points).
UPDRS - unified Parkinson's disease rating scale | 1.5-month Post-HIIT 1
  Motor and non-motor Parkinson's disease signs/symptoms will be evaluated using UPDRS (sections I - III, that include the items 1 -31). Each item is expressed in [points] from 0 to 4 points, with an interpretation that the higher value means the severe accentuation of sign/symptom. The total score will be reported, as the sum of the points of the sections I-III (the score in the range 0 - 176 points) and each section's score will be reported as well, i.e.: the sum of the points of the section I (sum of points for items 1-4 in the range 0 - 16 points), the sum of the points of the section II (sum of points for items 5-17 in the range 0 - 52 points), the sum of the points of the section III (sum of points for items 18-31 in the range 0 - 108 points).
UPDRS - unified Parkinson's disease rating scale | 3-months Post-HIIT 1
  Motor and non-motor Parkinson's disease signs/symptoms will be evaluated using UPDRS (sections I - III, that include the items 1 -31). Each item is expressed in [points] from 0 to 4 points, with an interpretation that the higher value means the severe accentuation of sign/symptom. The total score will be reported, as the sum of the points of the sections I-III (the score in the range 0 - 176 points) and each section's score will be reported as well, i.e.: the sum of the points of the section I (sum of points for items 1-4 in the range 0 - 16 points), the sum of the points of the section II (sum of points for items 5-17 in the range 0 - 52 points), the sum of the points of the section III (sum of points for items 18-31 in the range 0 - 108 points).
UPDRS - unified Parkinson's disease rating scale | 1-week Post-HIIT 2
  Motor and non-motor Parkinson's disease signs/symptoms will be evaluated using UPDRS (sections I - III, that include the items 1 -31). Each item is expressed in [points] from 0 to 4 points, with an interpretation that the higher value means the severe accentuation of sign/symptom. The total score will be reported, as the sum of the points of the sections I-III (the score in the range 0 - 176 points) and each section's score will be reported as well, i.e.: the sum of the points of the section I (sum of points for items 1-4 in the range 0 - 16 points), the sum of the points of the section II (sum of points for items 5-17 in the range 0 - 52 points), the sum of the points of the section III (sum of points for items 18-31 in the range 0 - 108 points).
UPDRS - unified Parkinson's disease rating scale | 1.5-month Post-HIIT 2
  Motor and non-motor Parkinson's disease signs/symptoms will be evaluated using UPDRS (sections I - III, that include the items 1 -31). Each item is expressed in [points] from 0 to 4 points, with an interpretation that the higher value means the severe accentuation of sign/symptom. The total score will be reported, as the sum of the points of the sections I-III (the score in the range 0 - 176 points) and each section's score will be reported as well, i.e.: the sum of the points of the section I (sum of points for items 1-4 in the range 0 - 16 points), the sum of the points of the section II (sum of points for items 5-17 in the range 0 - 52 points), the sum of the points of the section III (sum of points for items 18-31 in the range 0 - 108 points).
UPDRS - unified Parkinson's disease rating scale | 3-months Post-HIIT 2
  Motor and non-motor Parkinson's disease signs/symptoms will be evaluated using UPDRS (sections I - III, that include the items 1 -31). Each item is expressed in [points] from 0 to 4 points, with an interpretation that the higher value means the severe accentuation of sign/symptom. The total score will be reported, as the sum of the points of the sections I-III (the score in the range 0 - 176 points) and each section's score will be reported as well, i.e.: the sum of the points of the section I (sum of points for items 1-4 in the range 0 - 16 points), the sum of the points of the section II (sum of points for items 5-17 in the range 0 - 52 points), the sum of the points of the section III (sum of points for items 18-31 in the range 0 - 108 points).
BDNF - brain derived neurotrophic factor | Pre-HIIT 1 - it means up to 1-week before the HIIT 1 starts
  BDNF secretion level in blood expressed in [pg/mL]
BDNF - brain derived neurotrophic factor | 1-week Post-HIIT 1
  BDNF secretion level in blood expressed in [pg/mL]
BDNF - brain derived neurotrophic factor | 1.5-month Post-HIIT 1
  BDNF secretion level in blood expressed in [pg/mL]
BDNF - brain derived neurotrophic factor | 3-months Post-HIIT 1
  BDNF secretion level in blood expressed in [pg/mL]
BDNF - brain derived neurotrophic factor | 1-week Post-HIIT 2
  BDNF secretion level in blood expressed in [pg/mL]
BDNF - brain derived neurotrophic factor | 1.5-month Post-HIIT 2
  BDNF secretion level in blood expressed in [pg/mL]
BDNF - brain derived neurotrophic factor | 3-months Post-HIIT 2
  BDNF secretion level in blood expressed in [pg/mL]
NGF - nerve growth factor | Pre-HIIT 1 - it means up to 1-week before the HIIT 1 starts
  NGF secretion level in blood expressed in [pg/mL]
NGF - nerve growth factor | 1-week Post-HIIT 1
  NGF secretion level in blood expressed in [pg/mL]
NGF - nerve growth factor | 1.5-month Post-HIIT 1
  NGF secretion level in blood expressed in [pg/mL]
NGF - nerve growth factor | 3-months Post-HIIT 1
  NGF secretion level in blood expressed in [pg/mL]
NGF - nerve growth factor | 1-week Post-HIIT 2
  NGF secretion level in blood expressed in [pg/mL]
NGF - nerve growth factor | 1.5-month Post-HIIT 2
  NGF secretion level in blood expressed in [pg/mL]
NGF - nerve growth factor | 3-months Post-HIIT 2
  NGF secretion level in blood expressed in [pg/mL]
IGF 1 - insulin-like growth factor 1 | Pre-HIIT 1 - it means up to 1-week before the HIIT 1 starts
  IGF 1 secretion level in blood expressed in [pg/mL]
IGF 1 - insulin-like growth factor 1 | 1-week Post-HIIT 1
  IGF 1 secretion level in blood expressed in [pg/mL]
IGF 1 - insulin-like growth factor 1 | 1.5-month Post-HIIT 1
  IGF 1 secretion level in blood expressed in [pg/mL]
IGF 1 - insulin-like growth factor 1 | 3-months Post-HIIT 1
  IGF 1 secretion level in blood expressed in [pg/mL]
IGF 1 - insulin-like growth factor 1 | 1-week Post-HIIT 2
  IGF 1 secretion level in blood expressed in [pg/mL]
IGF 1 - insulin-like growth factor 1 | 1.5-month Post-HIIT 2
  IGF 1 secretion level in blood expressed in [pg/mL]
IGF 1 - insulin-like growth factor 1 | 3-months Post-HIIT 2
  IGF 1 secretion level in blood expressed in [pg/mL]
Val66Met polymorphism of BDNF - genotyping of BDNF polymorphism | Pre-HIIT 1 - it means up to 1-week before the HIIT 1 starts
  The single nucleotide polymorphism (SNP) BDNF Val66Met variant (rs 6265) will be genotyped by using the TaqMan SNP genotyping assay. Thermal cycling and end-point PCR (polymerase chain reaction) analysis will be performed on the Rotor-Gene Q 5plex real-time PCR Cycler and will be analyzed by Q-Rex-software. Genotype of BDNF polymorphism will be expressed in percentge values [% of genotype].

SECONDARY OUTCOMES:
H&Y scale - Hoehn and Yahr scale | Pre-HIIT 1 - it means up to 1-week before the HIIT 1 starts
  Parkinson's disease stage evaluation using H&Y scale, expressed in [points] from 1 to 5 points. The modified version of the H&Y scale will be used, in which: the score 1 means - unilateral involvement only; the score 1.5 means - unilateral and axial involvement; the score 2 means - bilateral involvement without impairment of balance; the score 2.5 means - mild bilateral disease with recovery on pull test; the score 3 means - mild to moderate bilateral disease, some postural instability, physically independent; the score 4 means - severe disability, still able to walk or stand unassisted; the score 5 means - wheelchair bound or bedridden unless aided.
H&Y scale - Hoehn and Yahr scale | 1-week Post-HIIT 1
  Parkinson's disease stage evaluation using H&Y scale, expressed in [points] from 1 to 5 points. The modified version of the H&Y scale will be used, in which: the score 1 means - unilateral involvement only; the score 1.5 means - unilateral and axial involvement; the score 2 means - bilateral involvement without impairment of balance; the score 2.5 means - mild bilateral disease with recovery on pull test; the score 3 means - mild to moderate bilateral disease, some postural instability, physically independent; the score 4 means - severe disability, still able to walk or stand unassisted; the score 5 means - wheelchair bound or bedridden unless aided.
H&Y scale - Hoehn and Yahr scale | 1.5-month Post-HIIT 1
  Parkinson's disease stage evaluation using H&Y scale, expressed in [points] from 1 to 5 points. The modified version of the H&Y scale will be used, in which: the score 1 means - unilateral involvement only; the score 1.5 means - unilateral and axial involvement; the score 2 means - bilateral involvement without impairment of balance; the score 2.5 means - mild bilateral disease with recovery on pull test; the score 3 means - mild to moderate bilateral disease, some postural instability, physically independent; the score 4 means - severe disability, still able to walk or stand unassisted; the score 5 means - wheelchair bound or bedridden unless aided.
H&Y scale - Hoehn and Yahr scale | 3-months Post-HIIT 1
  Parkinson's disease stage evaluation using H&Y scale, expressed in [points] from 1 to 5 points. The modified version of the H&Y scale will be used, in which: the score 1 means - unilateral involvement only; the score 1.5 means - unilateral and axial involvement; the score 2 means - bilateral involvement without impairment of balance; the score 2.5 means - mild bilateral disease with recovery on pull test; the score 3 means - mild to moderate bilateral disease, some postural instability, physically independent; the score 4 means - severe disability, still able to walk or stand unassisted; the score 5 means - wheelchair bound or bedridden unless aided.
H&Y scale - Hoehn and Yahr scale | 1-week Post-HIIT 2
  Parkinson's disease stage evaluation using H&Y scale, expressed in [points] from 1 to 5 points. The modified version of the H&Y scale will be used, in which: the score 1 means - unilateral involvement only; the score 1.5 means - unilateral and axial involvement; the score 2 means - bilateral involvement without impairment of balance; the score 2.5 means - mild bilateral disease with recovery on pull test; the score 3 means - mild to moderate bilateral disease, some postural instability, physically independent; the score 4 means - severe disability, still able to walk or stand unassisted; the score 5 means - wheelchair bound or bedridden unless aided.
H&Y scale - Hoehn and Yahr scale | 1.5-month Post-HIIT 2
  Parkinson's disease stage evaluation using H&Y scale, expressed in [points] from 1 to 5 points. The modified version of the H&Y scale will be used, in which: the score 1 means - unilateral involvement only; the score 1.5 means - unilateral and axial involvement; the score 2 means - bilateral involvement without impairment of balance; the score 2.5 means - mild bilateral disease with recovery on pull test; the score 3 means - mild to moderate bilateral disease, some postural instability, physically independent; the score 4 means - severe disability, still able to walk or stand unassisted; the score 5 means - wheelchair bound or bedridden unless aided.
H&Y scale - Hoehn and Yahr scale | 3-months Post-HIIT 2
  Parkinson's disease stage evaluation using H&Y scale, expressed in [points] from 1 to 5 points. The modified version of the H&Y scale will be used, in which: the score 1 means - unilateral involvement only; the score 1.5 means - unilateral and axial involvement; the score 2 means - bilateral involvement without impairment of balance; the score 2.5 means - mild bilateral disease with recovery on pull test; the score 3 means - mild to moderate bilateral disease, some postural instability, physically independent; the score 4 means - severe disability, still able to walk or stand unassisted; the score 5 means - wheelchair bound or bedridden unless aided.
S&E DLA scale - Schwab and England Daily Living Activity Scale | Pre-HIIT 1 - it means up to 1-week before the HIIT 1 starts
  S&E DLA scale measure of daily function of Parkinson's disease patients, expressed in [%] from 100 to 0 % (with the higher % value as the better score). The 100% score means that the person is completely independent; able to do all chores without slowness, difficulty or impairment; essentially normal; unaware of any difficulty. The 0% score describes the person bedridden with the only vegetative functions such as swallowing; bladder and bowel functions are not functioning.
S&E DLA scale - Schwab and England Daily Living Activity Scale | 1-week Post-HIIT 1
  S&E DLA scale measure of daily function of Parkinson's disease patients, expressed in [%] from 100 to 0 % (with the higher % value as the better score). The 100% score means that the person is completely independent; able to do all chores without slowness, difficulty or impairment; essentially normal; unaware of any difficulty. The 0% score describes the person bedridden with the only vegetative functions such as swallowing; bladder and bowel functions are not functioning.
S&E DLA scale - Schwab and England Daily Living Activity Scale | 1.5-month Post-HIIT 1
  S&E DLA scale measure of daily function of Parkinson's disease patients, expressed in [%] from 100 to 0 % (with the higher % value as the better score). The 100% score means that the person is completely independent; able to do all chores without slowness, difficulty or impairment; essentially normal; unaware of any difficulty. The 0% score describes the person bedridden with the only vegetative functions such as swallowing; bladder and bowel functions are not functioning.
S&E DLA scale - Schwab and England Daily Living Activity Scale | 3-months Post-HIIT 1
  S&E DLA scale measure of daily function of Parkinson's disease patients, expressed in [%] from 100 to 0 % (with the higher % value as the better score). The 100% score means that the person is completely independent; able to do all chores without slowness, difficulty or impairment; essentially normal; unaware of any difficulty. The 0% score describes the person bedridden with the only vegetative functions such as swallowing; bladder and bowel functions are not functioning.
S&E DLA scale - Schwab and England Daily Living Activity Scale | 1-week Post-HIIT 2
  S&E DLA scale measure of daily function of Parkinson's disease patients, expressed in [%] from 100 to 0 % (with the higher % value as the better score). The 100% score means that the person is completely independent; able to do all chores without slowness, difficulty or impairment; essentially normal; unaware of any difficulty. The 0% score describes the person bedridden with the only vegetative functions such as swallowing; bladder and bowel functions are not functioning.
S&E DLA scale - Schwab and England Daily Living Activity Scale | 1.5-month Post-HIIT 2
  S&E DLA scale measure of daily function of Parkinson's disease patients, expressed in [%] from 100 to 0 % (with the higher % value as the better score). The 100% score means that the person is completely independent; able to do all chores without slowness, difficulty or impairment; essentially normal; unaware of any difficulty. The 0% score describes the person bedridden with the only vegetative functions such as swallowing; bladder and bowel functions are not functioning.
S&E DLA scale - Schwab and England Daily Living Activity Scale | 3-months Post-HIIT 2
  S&E DLA scale measure of daily function of Parkinson's disease patients, expressed in [%] from 100 to 0 % (with the higher % value as the better score). The 100% score means that the person is completely independent; able to do all chores without slowness, difficulty or impairment; essentially normal; unaware of any difficulty. The 0% score describes the person bedridden with the only vegetative functions such as swallowing; bladder and bowel functions are not functioning.
MMSE - Mini Mental State Examination | Pre-HIIT 1 - it means up to 1-week before the HIIT 1 starts
  MMSE will be used to to exclude the Parkinson's disease patients with cognitive impairment, expressed in [points]in the range from 0 to 30 points. It is an 11-question measure that tests five areas of cognitive function: orientation, registration, attention and calculation, recall, and language. A score of 23 or lower is indicative of cognitive impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Jaroslaw Marusiak, PhD, Principal Investigator — University School of Physical Education in Wroclaw, Wroclaw, Poland
Locations (1):
- University School of Physical Education in Wroclaw, Wroclaw, Lower Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No